CLINICAL TRIAL: NCT02094976
Title: Comparison of Intraabdominal Pressure and Respiratory Parameter Changes According to Positional Apparatus in the Prone Position
Brief Title: Comparison of Intraabdominal Pressure
Acronym: IAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IAP_protocol
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Prone Position
Keywords: Prone position; Intra-abdominal pressure; Respiratory system compliance; Jackson table; Wilson frame; Chest roll

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group C (Active Comparator): Group C means active comparator group which use chest rolls intraoperatively for prone position.
  Interventions: Device: Chest roll
- Group W (Active Comparator): Group W means experimental group which use Wilson frame intraoperatively for prone position.
  Interventions: Device: Wilson frame
- Group J (Experimental): Group J means experimental group which use Jackson surgical table intraoperatively for prone position.
  Interventions: Device: Jackson surgical table

INTERVENTIONS:
Device: Jackson surgical table — After standard total intravenous anesthesia using propofol and remifentanil continous infusion, patients were turned to the prone position on a Jackson table with two padded supports on each side. The supports were positioned under the lateral chest and at the iliac crest.
  Arms: Group J
Device: Wilson frame — After standard total intravenous anesthesia using propofol and remifentanil continous infusion, patients were turned to the prone position on a Wilson frame. The supports were positioned vertically from shoulder to iliac crest.
  Arms: Group W
Device: Chest roll — After standard total intravenous anesthesia using propofol and remifentanil continous infusion, patients were turned to the prone position on a chest roll. The supports were positioned vertically from shoulder to iliac crest.
  Arms: Group C

SUMMARY:
Increased intra-abdominal pressure(IAP) might influence on perioperative morbidity related to increased CVP, PVWP, SVR, PAP and decreased venous return and cardiac output. Prone position has been known to increase IAP. In clinical field, various apparatuses has developed to minimize IAP elevation during prone position operation.

In this study, we would compare the changes of IAP and respiratory system compliance according to positional apparatus in prone position.

DETAILED DESCRIPTION:
In clinical field, Wison frame, chest rolls and Jackson table have been widely used for prone position surgery. Among those apparatus, Jackson table has padded supports under the chest and pelvis, so that the abdomen can hang freely and prevent the abdominal compression. By reducing abdominal and thoracic pressure, Jackson table would reduce blood loss, and less effects on pulmonary mechanics. But few studies has known to compare IAP with other positioning apparatus such as Wilson frame or chest roll.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for prone positioned spinal surgery
* ASA Physical Status Classification System class I or II

Exclusion Criteria:

* Patients who did not agree
* BMI > 30kg/m2
* Patients who did not insert urinary foley catheter
* Patients who have COPD or emphysema
* Patients who have severe spine deformities such as scoliosis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
changes of Intraabdominal presure (IAP) | 5 minute after position change
  Compare IAP changes from supine to prone according to the positional apparatus : Wilson frame, Chestrolls and Jackson table

SECONDARY OUTCOMES:
Changes of IAP and total respiratory system comliance (Crs) accoridng to PEEP change | 1min after PEEP change
  Compare IAP and Crs according to PEEP changes in each group. PEEP applied 0,3,6 and 9 cm H2O and recoding was done at 1min after PEEP change.
  Total respiratory system compliance (Crs) = TV/(Pplat-PEEP)
changes of dead space ventilation after position change | 5 minute after prone position
  After genearal anesthetic induction, arterial blood gas analyssis (ABGA)was done at supine position. And then the position was changed to prone. 5minutes after prone position change, ABGA repeated, and calculated the dead space ventilation at each point.
  Dead space ventilation (Vd/Vt) = [PaCo2-PETCO2]/PaCo2
  Finally, we would compare changes of dead space ventilation after position change.
Hemodynamic change | 1min after PEEP change
  Check the hemodynamic changes according to PEEP change : 0,3,6 and 9 cmH2O

OTHER OUTCOMES:
Estimated blood loss (EBL) | intraoperatively
  Compare the EBL among the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Pyung Park, MD PhD, Study Director — Professor; Eugene Kim, MD, Principal Investigator — Clinical Instuctor
Locations (1):
- Seoul National University of Hospital, Seoul, South Korea